CLINICAL TRIAL: NCT02880007
Title: A Prospective Open Label Phase II Study to Optimize the Dose in 3D Pulsed Dose Rate Brachytherapy in Patients With Locally Advanced Cervical Cancer
Brief Title: Dose Optimization in 3D Pulsed Dose Rate Brachytherapy for Patients With Locally Advanced Cervical Cancer
Acronym: TRIDICOL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-A00235-34
Record Dates: First submitted 2016-08-10; First posted 2016-08-26 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Cervical Adenocarcinoma; Stage IB Cervical Cancer; Stage II Cervical Cancer; Stage III Cervical Cancer
Keywords: Pulsed dose-rate brachytherapy; 3D dosimetry; Prospective Studies; Radiotherapy Dosage; Uterine Cervical Neoplasms/radiotherapy; Brachytherapy/methods
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ARM A (Experimental): Dose Optimization in 3D Pulsed Dose Rate Brachytherapy
  Interventions: Radiation: External Beam Radiation Therapy; Radiation: PDR Brachytherapy; Drug: Cisplatin

INTERVENTIONS:
Radiation: External Beam Radiation Therapy — 45 Gy pelvis / 25 fr
  Other Names: EBRT
Radiation: PDR Brachytherapy — 1 puls/hour ; 12 Gy / day
Drug: Cisplatin — increase in dose to the target volume at high risk (85 to 90 Gy over 90% of its volume) and the intermediate target volume (60 Gy to 90 % of its volume) in 3D Pulsed Dose Rate Brachytherapy
  Other Names: CDDP

SUMMARY:
This prospective phase II trial study aims to optimize the increase in dose to the target volume at high risk (85 to 90 Gy over 90% of its volume) and the intermediate target volume (60 Gy to 90 % of its volume) in 3D Pulsed Dose Rate Brachytherapy in treating patients with locally advanced cervical cancer.

DETAILED DESCRIPTION:
* The causes of treatment failure and death in cervical cancer are still often linked to a local cancer progression
* The importance of local control for healing, than the cervix situation in the center of pelvis between bladder and rectum which are sensitive organs to irradiation justify the use of utero-vaginal brachytherapy
* This open label, multicenter, phase II study evaluates the benefit of increasing in dose to the target volume at high risk and the intermediate target volume in 3D Pulsed Dose Rate Brachytherapy in treating patients with locally advanced cervical cancer.
* Local control and tolerance are evaluated

ELIGIBILITY:
Inclusion Criteria:

* primitive cervical cancer
* adenocarcinoma histologically advanced
* IB2, II and III stage
* curative treatment
* indication of utero-vaginal brachytherapy with external radiotherapy
* non-metastatic tumor and life expectancy > 6 months
* patient informed and follow possible
* performance status ≤ 2
* unplanned surgery
* age ≥ 18 years old
* ability to provide written informed consent before the start of any study specific procedures

Exclusion Criteria:

* primitive endometrial cancer
* other diseases
* carcinoma in situ and stages ≤ B
* distant metastases
* history of pelvic irradiation or a first pelvic cancer
* contraindication to MRI
* history of subtotal or total hysterectomy
* pregnant or breast feeding females
* inability to support low dose rate continuous brachytherapy or pulsed flow
* person in emergencies
* person unable to give personally consent
* patient participating in another clinical research except in case of local recurrence or observational research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-06-06 (Actual); Primary Completion 2014-02-10 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Increase the local control rate | 24 months
  Increasing local control in two years (from 71.0% to 86.7%) will be achieved by increasing the dose to the target volume (CTV and CTV-HR-RI) measured dose volume histograms

SECONDARY OUTCOMES:
Maintain the cumulative rate grade III and IV complications below 6.5% | 24 months
Relationship between the doses delivered to the target volume and local control | 24 months
Relationship between the doses delivered to the critical organs and rate of grade III and IV complications | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: PEIFFERT Didier, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (9):
- France (9):
  - CHU de Besançon, Besançon
  - Institut Bergonié, Bordeaux
  - Centre Georges-François Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - Centre Val d'Aurelle, Montpellier
  - Centre Paul Strauss, Strasbourg
  - Centre Claudius Regaud, Toulouse
  - CHRU Tours - Hôpital Bretonneau, Tours
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No